CLINICAL TRIAL: NCT02410330
Title: Therapeutic Use of Ultrasound in Acute Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Nebraska (Other)
Responsible Party: Principal Investigator, Wilson Mathias Junior, Director Echocardiography Laboratory - Heart Institute, University of Sao Paulo General Hospital
Other Study IDs: SDC 3562/10/151
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Therapeutic ultrasound; Angiographic recanalization rate; Salvagability index; Sonothrombolysis
MeSH Terms: interventions — Ultrasonic Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group I: Patients with acute STEMI will receive intravenous infusion of microbubbles (3% Definity) with Therapeutic ultrasound with 20 usec: custom designed high mechanical index (MI) impulses at 4-20 usec and >1.0 MI designed for the 1.7 MHz S5-1 transducer while waiting for percutaneous coronary intervention. Treatment will continue after procedure untill complete a total of 60 minutes.
  Interventions: Procedure: Therapeutic ultrasound with 20 usec
- Group II: Patients with acute STEMI will receive intravenous infusion of microbubbles (3% Definity) with therapeutic ultrasound with repeated diagnostic high mechanical index impulses (all <2 usec pulse duration; MI=1.0) whenever very low MI perfusion imaging detected microbubbles within the microvasculature. Treatment will be applied while patient waits for percutaneous coronary intervention. Treatment will continue after procedure untill complete a total of 60 minutes.
  Interventions: Procedure: Repeated diagnostic high mechanical index
- Group III: Patients with acute STEMI will receive intravenous infusion of microbubbles (3% Definity) while few limited diagnostic high MI impulses (n<5 per patient) will be applied to assess myocardial perfusion before and after percutaneous coronary intervention (PCI).

INTERVENTIONS:
Procedure: Therapeutic ultrasound with 20 usec — A custom designed high mechanical index (MI) impulses at 4-20 usec and >1.0 mechanical index designed for the 1.7 MHz S5-1 transducer
  Groups: Group I
Procedure: Repeated diagnostic high mechanical index — Repeated diagnostic high mechanical index impulses (all <2 usec pulse duration; MI=1.0) whenever very low mechanical index perfusion imaging detected microbubbles within the microvasculature
  Groups: Group II

SUMMARY:
In acute coronary artery disease, pre-clinical studies have indicated that, during a continuous infusion of intravenous perfluorocarbon containing microbubbles, the ultrasonic power delivered from a diagnostic ultrasound transducer is capable of restoring microcirculatory flow and improving epicardial recanalization rates obtained by conventional therapy, a process known by Sonothrombolysis. The investigators proposed to examine the feasibility, safety and efficacy of such an ultrasound guided approach in 100 patients with ST segment elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
In acute coronary artery disease, pre-clinical studies have indicated that, during a continuous infusion of intravenous perfluorocarbon containing microbubbles, the ultrasonic power delivered from a diagnostic ultrasound transducer is capable of restoring microcirculatory flow and improving epicardial recanalization rates obtained by conventional therapy, a process known by Sonothrombolysis. Since both diagnostic ultrasound and intravenous infusions of microbubbles are a Class I indication to assess regional and global left ventricular function and risk area in patients with ST segment elevation myocardial infarction (STEMI). The investigators propose to examine the effectiveness of microvascular sonothrombolysis.

A total of 100 patients with acute STEMI will be randomized to receive diagnostic ultrasound guided high mechanical index (MI) impulses in different approaches applied within and outside the risk area during a continuous infusion of intravenous 3% Definity® or placebo. The different ultrasound regimens are: Group I - a custom designed high mechanical index (MI) impulses at 4-20 usec and >1.0 MI designed for the 1.7 MHz S5-1 transducer; Group II - repeated diagnostic high MI impulses (all <2 usec pulse duration; MI=1.0 whenever very low MI perfusion imaging detected microbubbles within the microvasculature; Group III (control), where a few limited diagnostic high MI impulses (n<5 per patient) will be applied to assess myocadial perfusion before and after percutaneous coronary intervention (PCI). All patients will receive the conventional PCI approach, including 325 milligrams Aspirin, 600 milligrams Clopidogrel, and heparin bolus (5000 units), followed by primary PCI using glycoprotein 2b/3a inhibitors as anti-thrombotic agents using established protocols. Besides angiographic recanalization rates at the time of presentation to the catheterization laboratory, the patients will have a magnetic resonance exam performed at 72-96 hours post infarcton to quantify the myocardial salvagability index. Quantitative assessments of ejection fraction will be made at this time as well.Overall survival (OS), defined as the time from the start of treatment to death from any cause, will be evaluated.Comparisons between the three groups will be made on door to dilation times, survival, angiographic recanalization rates (ARR) at initial angiography, and reduction in infarct size determined by the salvagability index (SI) at magnetic resonance imaging 72-96 hours post STEMI. Left ventricular function and perfusion parameters by echocardiography will also be evaluated during, at 72-96 hours and at 6 months in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥30 years with STEMI with less than 12 hours of chest pain onset.
* Eligible for emergent PCI therapy.
* No contraindications or hypersensitivities to ultrasound contrast agents

Exclusion Criteria:

* Known or suspected hypersensitivity to ultrasound contrast agent used for the study.
* Cardiogenic Shock.
* Life expectancy of less than two months or terminally ill.
* Known bleeding diathesis or contraindication to glycoprotein 2b/3a inhibitors, anticoagulants, or aspirin.
* Known large right to left intracardiac shunts or severe pulmonary hypertension.
* Patients who received thrombolytic therapy previously to enrollment.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute ST elevation myocardial infarction (STEMI) with less than 12 hours of chest pain onset, eligible for emergent percutaneous coronary intervention therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Angiographic recanalization rate | At initial angiography
  Percentage of patients with acute STEMI and open artery at initial angiography (TIMI I)

SECONDARY OUTCOMES:
Salvagability index | 72-96 hours post infarction
  Percentage of myocardium with viability within the risk area obtained by magnetic ressonance imaging
Overall survival | 30 days post infarction
  The time from the start of treatment to death from any cause
Left ventricular function and perfusion parameters | 72-96 hours and at 6 months
  left ventricular volumes, ejection fraction, longitudinal strain, diastolic function and infarct size by myocardial contrast echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Mathias Jr, MD, Principal Investigator — Heart Institute - University of São Paulo Medical School
Locations (1):
- Heart Institute (InCor), São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mathias W Jr, Tsutsui JM, Tavares BG, Fava AM, Aguiar MOD, Borges BC, Oliveira MT Jr, Soeiro A, Nicolau JC, Ribeiro HB, Chiang HP, Sbano JCN, Morad A, Goldsweig A, Rochitte CE, Lopes BBC, Ramirez JAF, Kalil Filho R, Porter TR; MRUSMI Investigators. Sonothrombolysis in ST-Segment Elevation Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention. J Am Coll Cardiol. 2019 Jun 11;73(22):2832-2842. doi: 10.1016/j.jacc.2019.03.006. Epub 2019 Mar 17. PMID 30894317
- [Result] Aguiar MOD, Tavares BG, Tsutsui JM, Fava AM, Borges BC, Oliveira MT Jr, Soeiro A, Nicolau JC, Ribeiro HB, Chiang HP, Sbano JCN, Goldsweig A, Rochitte CE, Lopes BBC, Ramirez JAF, Kalil Filho R, Porter TR, Mathias W Jr. Sonothrombolysis Improves Myocardial Dynamics and Microvascular Obstruction Preventing Left Ventricular Remodeling in Patients With ST Elevation Myocardial Infarction. Circ Cardiovasc Imaging. 2020 Apr;13(4):e009536. doi: 10.1161/CIRCIMAGING.119.009536. Epub 2020 Apr 21. PMID 32312114
- [Derived] Mathias W Jr, Tsutsui JM, Tavares BG, Xie F, Aguiar MO, Garcia DR, Oliveira MT Jr, Soeiro A, Nicolau JC, Lemos PA Neto, Rochitte CE, Ramires JA, Kalil R Filho, Porter TR. Diagnostic Ultrasound Impulses Improve Microvascular Flow in Patients With STEMI Receiving Intravenous Microbubbles. J Am Coll Cardiol. 2016 May 31;67(21):2506-15. doi: 10.1016/j.jacc.2016.03.542. PMID 27230046